STATISTIC ANALYSIS

**Identifiers: NCT03636386** 

**Protocol ID: 60312069** 

Date of the document: August 15, 2019

Brief Title: Percutaneous Microelectrolysis on Myofascial

**Trigger Points Pain. (MEP)** 

Official Title: Effectiveness of Percutaneous Microelectrolysis in

the Decrease of Pain in Myofascial Trigger Points: Evaluation

Through Algometry and Visual Analog Scale. Randomized

**Controlled Trial.** 

Statistical analysis

The data collected from the participants were tabulated in a Microsoft Excel® program table,

and subsequently a mother base table was made with the data obtained after the intervention.

The STATA® v.13 program was used for statistical analysis, where the proposed variables

were analyzed; Painful pressure threshold (UPD) and pain intensity (ID) as primary variables,

and sex, body mass index, shortened trapezius laterality, spiny-acromion process distance as

secondary variables.

Statistical analysis began by comparing both study groups (microelectrolysis, n = 30 and

control, n = 24). The Shapiro-Wilk test was applied to determine the use of parametric or

non-parametric tests. The analysis of the pain pressure threshold (UPD) and pain intensity

(ID) variables before intervention and the secondary variables sex, body mass index (BMI)

and laterality (shortened trapezoid), spiny process-acromion distance (cm) being obtained a

normal distribution behavior except for the spiny process-acromion process variable (p value

1

<0.05). The variables UPD (Kg / cm<sup>2</sup>), Intensity (millimeters) and BMI (Kg / m2) were analyzed with the T-Student test (T-Test) showing that there are no statistically significant

differences between the microelectrolysis (MEP) and control group (p value> 0.05). On the other hand, for the analysis of the sex variable, the chi-square test (x2) was used, showing no differences between the study groups (p value> 0.05). For the laterality variable (presence of trigger point on the right and left side), Fisher's statistical test (F-Fisher) was used, not showing significant differences between the groups (p value> 0.05). For the spiny process-acromion process variable, given the result of the S-Wilk test, the U-Mann Whitney test was used, neither showing a difference between the groups (p value> 0.05). This analysis allowed to determine the homogeneity of both groups to enhance the interventions, MEP and conventional ultrasound for the experimental group, and only ultrasound for the control group (Table 1. Characterization of study groups).

#### Results

Sample was categorized in relation age, sex, BMI, SUTL, PPT and PI preintervention (PPTpre and PIpre). S-Wilk test was applied to analyze normal distribution and then compare homogeneity between groups (Table 1. Characterization of study groups). Statistical analysis performed in relation primary and second variables not shown statistically differences, so groups are comparable at beginning of study.

| Variable | MEP<br>(n = 24) | Control<br>(n = 24) | p-value | Sample distribution |
|---|---|---|---|---|
| sex (%)<br>men<br>women | 11 (22,9%)<br>13 (27,1%) | 12 (25,0%)<br>12 (25,0%) | <i>p</i> = 0,7730* | Normal* |
| Age (mean,+/-DS) | 22,5+/-1,9 | 22,0+/-1,6 | p = 0,2993** | Normal** |

| BMI (Kg/m2)<br>(mean +/-DS) | 24,5 +/- 3,4 | 22,9+/-2,3 | p =0,0616** | Normal** |
|---|---|---|---|---|
| Short trapezius<br>muscle laterality (%)<br>right<br>left | 17 (70,8%)<br>7 (29,2%) | 20 (83,3%)<br>4 (16,7%) | p = 0,2470*** | Normal*** |
| SP-AC distance (cm) (mean+/-DS) | 9,2+/-1,8 | 8,4+/-1,7 | p = 0,1241** | Normal** |
| PPTpre 1 (Kg/cm2)<br>(mean +/-DS) | 1,4+/-0,2 | 1,4+/-0,2 | <i>p</i> = 0,5734** | Normal** |
| PIpre1 (mm)<br>(mean +/- DS) | 32,1+/-13,6 | 31.4 +/- 15.1 | p = 0,8729** | Normal** |

**Table 1. Characterization of study groups.** Variable sex and short trapezius muscle laterality is represented in frequencies (%). Values for continuous variables are in means with their corresponding standard deviation (DS). Variable sex was analyzed using xi2 test\*. For the analysis of continuous variables, the T-Student test was used\*\*. Variable short trapezius laterality was analyzed with the F-Fisher test\*\*\*.

BMI: body mass index, SUTL: short upper trapezius muscle laterality, SP-AC distance: distance spinous process from C7 to acromion, PPTpre: pain pressure threshold pre intervention at day one, PIpre: pain intensity pre intervention at day one. p > 0.05\*\*\*\*

Table 2 shows evaluation results obtained for PPTpre, PPTpost, PPT2, PPT3, PPTdiff1-1, PPTdiff2-1, PPTdiff3-1, PIpre, PIpost, PI2, PI3, PIdiff1-1, PIdiff2-1 and PIdiff3-1 represented for each group. Averages with respective standard deviations (SD) were determined for all variables. S-Wilk showed a normal distribution, so T-Student test was used. PPTdiff1-1 for MEP group was 0,2+/-0,2 and control 0,2+/-0,2 without statistical difference between groups (p=0,0520). Means for PPTdiff2-1 for MEP group was 0,4+/-2 and control 0,2+/-0,2 showing statistically significant differences in favor of the experimental group (p=0,0032\*). Means for PPTdiff3-1 for MEP group was 0,5+/-0,4 and control 0,3+/-0,3 without difference between groups (p=0,0548). PIdiff1-1 for MEP group was -7,5+/-8,4 and control -6,6+/-8,6 without statistical difference between groups (p=0,3557). Means for PIdiff2-1 for MEP group was -10,5+/-11,9 and control -7,6+/-12,1 without statistically differences (p=0,2055). Means for PPTdiff3-1 for MEP group was -14+/-12,3 and control -11,5+/-13,1 without difference between groups (p=0,2457).

| Variable | Experimental (n = 24) | Control (n = 24) | p-value | Variable | Experimental (n = 24) | Control (n = 24) | p-value |
|---|---|---|---|---|---|---|---|
| PPTpre (Kg/cm²)<br>(mean +/-DS) | 1,4+/-0,2 | 1,4+/-0,2 | p = 0,6299 | PIpre (mm)<br>(mean +/-DS) | 32,1+/-13,6 | 31.4 +/-<br>15.1 | p = 0,8729 |
| PPTpost (Kg/cm²)<br>(mean +/-DS) | 1,6+/-0,2 | 1,6+/-0,2 | p = 0,4008 | PIpost (mm)<br>(mean +/-DS) | 24,6+/-12,7 | 24,8+/-<br>15,1 | p = 0,9508 |
| PPT2 (Kg/cm²)<br>(mean +/-DS) | 1,7 +/-0,1 | 1,6+/-0,2 | p = 0,0062* | PI2 (mm)<br>(mean +/-DS) | 21,6+/-11,0 | 23,8+/-<br>14,0 | p = 0,5461 |
| PPT3 (Kg/cm²)<br>(mean +/-DS) | 1,9 +/-0,3 | 1,7+/-0,2 | p = 0,0805 | PI3 (mm)<br>(mean +/-DS) | 18,1+/-9,9 | 20,0+/-<br>13,2 | p = 0,5815 |
| PPTdiff1-1 (Kg/cm²)<br>(mean +/-DS) | 0,2+/-0,2 | 0,2+/-0,1 | p = 0,0520 | PIdiff1-1 (mm)<br>(mean +/-DS) | -7,5+/-8,4 | -6,6+/-<br>8,6 | p = 0.3557 |
| PPTdiff2-1 (Kg/cm²)<br>(mean +/-DS) | 0,4+/-0,2 | 0,2+/-0,2 | p = 0,0032* | PIdiff2-1 (mm)<br>(mean +/-DS) | -10,5+/-11,9 | -7,6+/-<br>12,1 | p = 0,2055 |
| PPTdiff3-1 (Kg/cm²)<br>(mean +/-DS) | 0,5+/-0,4 | 0,3+/-0,3 | p = 0,0548 | PIdiff3-1 (mm)<br>(mean +/-DS) | -14,0+/-12,3 | -11,5+/-<br>13,1 | p = 0,2457 |

**Table 1. PPT, PI, PPTdiff and PIdiff variables measured by groups after baseline ultrasound treatment** and MEP intervention for all evaluation sessions. Values are means with their corresponding standard deviation (SD). Data analyzed using parametric T-Student test to compare intergroup differences for variables. PPT1-1: pain pressure threshold difference pre and postintervention at day one, PPT2-1: pain pressure threshold difference preintervention at day one and second evaluation at day tree, PPT3-1: pain pressure threshold difference pre intervention at day one and third evaluation at day seven. PIdiff1-1: pain intensity pre and post intervention at day one, PI2-1: pain intensity preintervention at day one and second evaluation at day tree, PI3-1: pain intensity difference preintervention at day one and third evaluation at day seven. \*p < 0.05.

Table 3 shows the PPTdiff and PIdiff between days one, three and seven obtained for MEP group. S-Wilk showed a normal distribution, so T-Student test was used. Significant differences are observed in MEP group for PPTdiff1-1 (p=0,0000), PPTdiff2-1 (p=0,0000), PPTdiff3-1 (p=0,0000), PIdiff1-1 (p=0,0001), PIdiff2-1 (p=0,0001) and PIdiff3-1 (p=0,0008). There are also statistically significant differences for control group in the variables PPTdiff1-1 (p=0.0001), PPTdiff2-1 (p=0.0001), PPTdiff3-1 (p=0,0002), PIdiff1-1 (p=0,0008) and PIdiff3-1 (p=0.0001).

| Variable | Experimental (n = 24) | p-value | Control (n = 30) | p-value |
|---|---|---|---|---|
| PPTdiff1-1 (Kg/cm²)<br>(mean +/-DS) | 0,2+/-0,2 | p = 0,0000* | 0,2+/-0,1 | <i>p</i> = 0,0001* |
| PPTdiff2-1 (Kg/cm²)<br>(mean +/-DS) | 0,4+/-0,2 | p = 0,0000* | 0,2+/-0,2 | p = 0,0000* |
| PPTdiff3-1 (Kg/cm²)<br>(mean +/-DS) | 0,5+/-0,4 | p = 0,0000* | 0,3+/-0,3 | <i>p</i> = 0,0002* |
| PIdiff1-1 (mm)<br>(mean +/-DS) | -8,0+/-8,6 | p = 0,0001* | -6,6+/-8,6 | p = 0,0022* |
| PIdiff2-1 (mm)<br>(mean +/-DS) | -10,8+/-12,2 | p = 0,0001* | -7,6+/-12,1 | p = 0,0008* |
| PIdiff3-1 (mm)<br>(mean +/-DS) | -14,3+/-14,5 | p = 0,0008* | -11,5+/-13,1 | p = 0,0001* |

Table 3. Description of PPT, PI, PPTdiff and PIdiff variables measured by groups after baseline ultrasound treatment and MEP intervention for all evaluation sessions. Values are means with their corresponding standard deviation (SD). Data analyzed using parametric T-Student test to compare intragroup differences for PPT and PI differences. Statistically significant difference for each variable was shown when groups were analyzed individually. \*p < 0.05.

Figure 1 represents PPT, PPTdiff, PI and PIdiff for sessions one, three and seven for groups. Statistically significant differences are seen in the second evaluation session between MEP and control group. In both groups are significant differences for PPTdiff and PIdiff when they are analyzed independently, visualizing an improvement pressure tolerance and decrease in pain intensity between evaluation sessions.



13.0 Copyright 1985-2013 StataCorp LP Statistics/Data Analysis StataCorp 4905 Lakeway Drive Special Edition College Station, Texas 77845 USA 800-STATA-PC http://www.stata.com 979-696-4600 stata@stata.com 979-696-4601 (fax) 3-user Stata network perpetual license: Serial number: 501306208483 Licensed to: IDRE-UCLA IDRE-UCLA Notes: 1. (-set maxvar-) 5000 maximum variables use "/Users/jaimeopazoc/Documents/UNAB/BASES/DLB2018/DIC2018/121218.dta" . sum edadaos Variable | Obs Mean Std. Dev. Max edadaos | 54 22.12963 1.770261 19 28 . swilk edadaos Shapiro-Wilk W test for normal data Variable | Obs Prob>z

0.04955

edadaos | 54 0.95679 2.159 1.649

| . bysort grupo:s | | daos<br> | | | |
|---|---|---|---|---|---|
| grupo = MEP | | | | | |
| | Shapiı | o-Wilk W te | st for no | rmal data | |
| Variable <br> | | | | | |
| edadaos | 30 | 0.91504 | 2.700 | 2.054 | 0.01999 |
| > grupo = CONTR | | | | | |
| | Shapiı | o-wilk w te | st for no | rmal data | |
| Variable <br> | | | | | |
| edadaos | | | | | |
| . (la edad no se<br>unrecognized com<br>r(199);<br>. h tabstat | | | _ | O MEP) | |
| bysort grupo:t | abstat ed | dadaos, s(me | ed iqr) | | |
| variable | p50 | iqr | | | |
| | 22 | 2 | | | |

| variable | p50 | iqr |
|----------|-----|-----|
| edadaos | 22 | 2.5 |

. bysort grupo:sum edadaos,detail

-----

-> grupo = MEP

# Edad (años)

| | Percentiles | Smallest | | |
|-----|-------------|----------|-------------|----------|
| 1% | 19 | 19 | | |
| 5% | 20 | 20 | | |
| 10% | 21 | 21 | Obs | 30 |
| 25% | 21 | 21 | Sum of Wgt. | 30 |
| 50% | 22 | | Mean | 22.26667 |
| | | Largest | Std. Dev. | 1.892514 |
| 75% | 23 | 24 | | |
| 90% | 24.5 | 25 | Variance | 3.581609 |
| 95% | 27 | 27 | Skewness | 1.316004 |
| 99% | 28 | 28 | Kurtosis | 5.056147 |

\_\_\_\_\_

-> grupo = CONTROL

## Edad (años)

| | Percentiles | Smallest | | |
|-----|-------------|----------|-------------|----------|
| 1% | 19 | 19 | | |
| 5% | 19 | 19 | | |
| 10% | 20 | 20 | Obs | 24 |
| 25% | 21 | 20 | Sum of Wgt. | 24 |
| 50% | 22 | | Mean | 21.95833 |
| | | Largest | Std. Dev. | 1.627993 |
| 75% | 23.5 | 24 | | |
| 90% | 24 | 24 | Variance | 2.650362 |

| 95% | 24 | 24 | Skewness | 1788824 |
|-----|----|----|----------|---------|
| 99% | 24 | 24 | Kurtosis | 1.92126 |

. ranksum edadaos, by( grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| expected | rank sum | obs | grupo |
|------------|------------|----------|------------------|
| 825<br>660 | 835<br>650 | 30<br>24 | MEP <br>CONTROL |
| 1485 | 1485 | <br>54 | combined |

unadjusted variance 3300.00 adjustment for ties -176.48 ------- adjusted variance 3123.52

Ho: edadaos(grupo==MEP) = edadaos(grupo==CONTROL)

z = 0.179Prob > |z| = 0.8580

. bysort grupo:swilk updpre1kgcm2 updpost1kgcm2 upd2kgcm2 updda3kgcm2 DELTAUPDPREPOST DELTAUPDDOSPRE DELTAUPDTRESPRE

-----

-----

-> grupo = MEP

### Shapiro-Wilk W test for normal data

| Variable | I | Obs | W | V | z | Prob>z |
|--------------|--------|-----|---------|-------|--------|---------|
| updpre1kgcm2 | -+<br> | 30 | 0.93435 | 2.087 | 1.521 | 0.06414 |
| updpost1kg~2 | | 30 | 0.97931 | 0.658 | -0.867 | 0.80690 |
| upd2kgcm2 | | 30 | 0.95820 | 1.329 | 0.588 | 0.27842 |
| updda3kgcm2 | | 30 | 0.79882 | 6.394 | 3.836 | 0.00006 |
| DELTAUPDPR~T | | 30 | 0.98513 | 0.473 | -1.549 | 0.93931 |
| DELTAUPDDO~E | | 30 | 0.96048 | 1.256 | 0.472 | 0.31863 |
| DELTAUPDTR~E | | 30 | 0.81101 | 6.007 | 3.707 | 0.00010 |

-----

-----

-> grupo = CONTROL

### Shapiro-Wilk W test for normal data

| Variable | Obs | W | V | z | Prob>z |
|--------------|-----|---------|-------|--------|---------|
| + | | | | | |
| updpre1kgcm2 | 24 | 0.95997 | 1.080 | 0.157 | 0.43781 |
| updpost1kg~2 | 24 | 0.95040 | 1.338 | 0.594 | 0.27640 |
| upd2kgcm2 | 24 | 0.95013 | 1.345 | 0.604 | 0.27278 |
| updda3kgcm2 | 24 | 0.83305 | 4.503 | 3.068 | 0.00108 |
| DELTAUPDPR~T | 24 | 0.98149 | 0.499 | -1.416 | 0.92169 |
| DELTAUPDDO~E | 24 | 0.96511 | 0.941 | -0.124 | 0.54934 |
| DELTAUPDTR~E | 24 | 0.95140 | 1.311 | 0.552 | 0.29044 |

. bysort grupo:sum updpre1kgcm2 updpost1kgcm2 upd2kgcm2 updda3kgcm2
DELTAUPDPREPOST DELTAUPDDOSPRE DELTAUPDTRESPRE, d
> etail

-----

-----

-> grupo = MEP

## UPD PRE 1 (Kg/cm2)

| | Percentiles | smallest | | |
|-----|-------------|----------|-------------|----------|
| 1% | 1.1 | 1.1 | | |
| 5% | 1.15 | 1.15 | | |
| 10% | 1.2 | 1.2 | Obs | 30 |
| 25% | 1.25 | 1.2 | Sum of Wgt. | 30 |
| 50% | 1.4 | | Mean | 1.419333 |
| | | Largest | Std. Dev. | .200309 |
| 75% | 1.61 | 1.72 | | |
| 90% | 1.725 | 1.73 | Variance | .0401237 |
| 95% | 1.75 | 1.75 | Skewness | .3370372 |
| 99% | 1.77 | 1.77 | Kurtosis | 1.843133 |

#### UPD POST 1 (Kg/cm2)

-----

Percentiles Smallest 1% 1.2 1.2

| 5% | 1.21 | 1.21 | | |
|-------|-------------|-----------------------|--------------|----------|
| 10% | 1.35 | 1.3 | Obs | 30 |
| 25% | 1.5 | 1.4 | Sum of Wgt. | 30 |
| 50% | 1.61 | | Mean | 1.6 |
| | | Largest | Std. Dev. | .1863811 |
| 75% | 1.73 | 1.8 | | |
| 90% | 1.81 | 1.82 | Variance | .0347379 |
| 95% | 1.92 | 1.92 | Skewness | 3238814 |
| 99% | 1.95 | 1.95 | Kurtosis | 2.769574 |
| | | UPD 2 (Kg/cn | | |
| | Percentiles | <br>Smallest | | |
| 1% | 1.45 | 1.45 | | |
| 5% | 1.49 | 1.49 | | |
| 10% | 1.51 | 1.5 | Obs | 30 |
| 25% | 1.63 | 1.52 | Sum of Wgt. | 30 |
| Z J/0 | 1.03 | 1.32 | Juli Of Wgc. | 30 |
| 50% | 1.705 | | Mean | 1.713 |
| | | Largest | Std. Dev. | .1366382 |
| 75% | 1.82 | 1.9 | | |
| 90% | 1.9 | 1.9 | Variance | .01867 |
| 95% | 1.9 | 1.9 | Skewness | 1850884 |
| 99% | 1.93 | 1.93 | Kurtosis | 2.131007 |
| | | upp día 2 (va | (cm2) | |
| | | UPD día 3 (Kg/<br> | · CIII2 ) | |
| | Percentiles | Smallest | | |
| 1% | 1.35 | 1.35 | | |
| 5% | 1.52 | 1.52 | | |
| 10% | 1.605 | 1.6 | Obs | 30 |
| 25% | 1.65 | 1.61 | Sum of Wgt. | 30 |
| F.00/ | 1 70 | | | 1 022 |
| 50% | 1.78 | | Mean | 1.822 |
| | | Largest | Std. Dev. | .2699221 |
| 75% | 1.85 | 2 | | |
| 90% | 2.075 | 2.15 | Variance | .0728579 |
| 95% | 2.6 | 2.6 | Skewness | 1.807479 |
| 99% | 2.7 | 2.7 | Kurtosis | 6.988866 |
| | | DELTAUPDPREF | POST | |
| | | ·•· - · ·· <b>-</b> · | | |

| | Percentiles | Smallest | | |
|-----|-------------|--------------|-------------|-----------|
| 1% | 1999999 | 1999999 | | |
| 5% | 1800001 | 1800001 | | |
| 10% | 095 | 12 | Obs | 30 |
| 25% | .0500001 | 0699999 | Sum of Wgt. | 30 |
| 50% | .17 | | Mean | .1806667 |
| | | Largest | Std. Dev. | .208044 |
| 75% | .34 | .4299999 | | |
| 90% | .46 | .49 | Variance | .0432823 |
| 95% | .55 | .55 | Skewness | .1213796 |
| 99% | . 5999999 | .5999999 | Kurtosis | 2.355019 |
| | | DELTAUPDDOS | PRE | |
| | Percentiles | | | |
| 1% | 09 | 09 | | |
| 5% | 0400001 | 0400001 | | |
| 10% | 03 | 03 | Obs | 30 |
| 25% | .1 | 03 | Sum of Wgt. | 30 |
| 50% | . 3 | | Mean | . 2936667 |
| | | Largest | Std. Dev. | .2249978 |
| 75% | .4899999 | .5500001 | | |
| 90% | .575 | .5999999 | Variance | .050624 |
| 95% | .64 | .64 | Skewness | 0390176 |
| 99% | . 6999999 | .6999999 | Kurtosis | 1.852427 |
| | | DELTAUPDTRES | SPRE | |
| | Percentiles | Smallest | | |
| 1% | .02 | .02 | | |
| 5% | .03 | .03 | | |
| 10% | .045 | .03 | Obs | 30 |
| 25% | .13 | .0600001 | Sum of Wgt. | 30 |
| 50% | .335 | | Mean | .4026667 |
| | | Largest | Std. Dev. | .3711764 |
| 75% | .52 | .65 | | |
| 90% | .8 | .95 | Variance | .1377719 |
| 95% | 1.4 | 1.4 | Skewness | 1.752146 |
| 99% | 1.6 | 1.6 | Kurtosis | 6.121863 |

-----

\_\_\_\_\_\_

## -> grupo = CONTROL

# UPD PRE 1 (Kg/cm2)

| | | PRE 1 (Rg/ | | |
|----------|--------------|---------------|--------------------|----------|
| | Percentiles | Smallest | | |
| 1% | 1 | 1 | | |
| 5% | 1.1 | 1.1 | | |
| 10% | 1.15 | 1.15 | Obs | 24 |
| 25% | 1.26 | 1.2 | Sum of Wgt. | 24 |
| 50% | 1.335 | | Mean | 1.4 |
| | | Largest | Std. Dev. | .2151036 |
| 75% | 1.59 | 1.69 | | |
| 90% | 1.7 | 1.7 | Variance | .0462696 |
| 95% | 1.71 | 1.71 | Skewness | .2114386 |
| 99% | 1.8 | 1.8 | Kurtosis | 2.093726 |
| | | UPD POST 1 (K | | |
| | Percentiles | Smallest | | |
| 1% | 1.1 | 1.1 | | |
| 5% | 1.21 | 1.21 | | |
| 10% | 1.32 | 1.32 | Obs | 24 |
| 25% | 1.425 | 1.35 | Sum of Wgt. | 24 |
| 50% | 1.6 | | Mean | 1.56 |
| | | Largest | Std. Dev. | .1901029 |
| 75% | 1.71 | 1.73 | | |
| 90% | 1.8 | 1.8 | Variance | .0361391 |
| 95% | 1.81 | 1.81 | Skewness | 6924839 |
| 99% | 1.83 | 1.83 | Kurtosis | 2.854815 |
| | | UPD 2 (Kg/cr | n2) | |
| | Percentiles | Smallest | | |
| | | 1.31 | | |
| 1% | 1.31 | 1.51 | | |
| 1%<br>5% | 1.31<br>1.35 | 1.35 | | |
| | | | Obs | 24 |
| 5% | 1.35 | 1.35 | Obs<br>Sum of Wgt. | 24<br>24 |

| | | Largest | Std. Dev. | .1578111 |
|------|-------------|----------------|-------------|------------|
| 75% | 1.74 | 1.77 | | |
| 90% | 1.8 | 1.8 | Variance | .0249043 |
| 95% | 1.8 | 1.8 | Skewness | 423535 |
| 99% | 1.88 | 1.88 | Kurtosis | 2.272104 |
| | | UPD día 3 (Kg/ | /cm2) | |
| | Percentiles | Smallest | | |
| 1% | 1.42 | 1.42 | | |
| 5% | 1.43 | 1.43 | | |
| 10% | 1.55 | 1.55 | Obs | 24 |
| 25% | 1.645 | 1.6 | Sum of Wgt. | 24 |
| 50% | 1.7 | | Mean | 1.72375 |
| 30% | 1.7 | Largest | Std. Dev. | .1880752 |
| 75% | 1.805 | 1.85 | Stu. Dev. | . 10007 32 |
| 90% | 1.85 | 1.85 | Variance | .0353723 |
| 95% | 1.92 | 1.92 | Skewness | 1.734271 |
| 99% | 2.4 | 2.4 | Kurtosis | 8.292314 |
| 33/0 | 2.4 | 2.4 | Rui COSTS | 0.292314 |
| | | DELTAUPDPREF | POST | |
| | Percentiles | <br>Smallest | | |
| 1% | 14 | 14 | | |
| 5% | 01 | 01 | | |
| 10% | 0 | 0 | Obs | 24 |
| 25% | .045 | 0 | Sum of Wgt. | 24 |
| 50% | .135 | | Mean | .16 |
| | | Largest | Std. Dev. | .1498405 |
| 75% | . 265 | .3200001 | | |
| 90% | .34 | .34 | Variance | .0224522 |
| 95% | .4 | .4 | Skewness | .3053529 |
| 99% | .5 | .5 | Kurtosis | 2.734097 |
| | | DELTAUPDDOSF | PRE<br> | |
| | Percentiles | Smallest | | |
| 1% | 2199999 | 2199999 | | |
| 5% | 08 | 08 | | |
| 10% | .02 | .02 | Obs | 24 |
| 25% | .105 | .09 | Sum of Wgt. | 24 |
| 23/0 | | | | |

| 50% | .19 | | Mean | .215 |
|-----|-------------|--------------|-------------|----------|
| | | Largest | Std. Dev. | .1936604 |
| 75% | .29 | .4000001 | | |
| 90% | .48 | .48 | Variance | .0375043 |
| 95% | .54 | .54 | Skewness | .3329579 |
| 99% | . 6999999 | . 6999999 | Kurtosis | 3.825891 |
| | | DELTAUPDTRES | SPRE | |
| | | | -<br> | |
| | Percentiles | Smallest | | |
| 1% | 1999999 | 1999999 | | |
| 5% | 1 | 1 | | |
| 10% | 0100001 | 0100001 | Obs | 24 |
| 25% | .145 | 0 | Sum of Wgt. | 24 |
| 50% | .3099999 | | Mean | .32375 |
| | | Largest | Std. Dev. | .3024798 |
| 75% | .43 | .7199999 | | |
| 90% | .73 | .73 | Variance | .091494 |
| 95% | .75 | .75 | Skewness | .7723583 |
| 99% | 1.16 | 1.16 | Kurtosis | 3.854242 |

. bysort grupo:ranksum updpre1kgcm2 updpost1kgcm2 upd2kgcm2 updda3kgcm2
DELTAUPDPREPOST DELTAUPDDOSPRE DELTAUPDTRESPR
> E, detail

\_\_\_\_\_

\_\_\_\_\_

-> grupo = MEP
too many variables specified
r(103);

. ranksum updpre1kgcm2, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| grupo | l obs | rank sum | expected |
|---------|-------|----------|----------|
| MEP | • | 840 | 825 |
| CONTROL | | 645 | 660 |

combined | 54 1485 1485

unadjusted variance 3300.00 adjustment for ties -3.77 ------ adjusted variance 3296.23

Ho: updpre~2(grupo==MEP) = updpre~2(grupo==CONTROL)

z = 0.261Prob > |z| = 0.7939

. ranksum updpost1kgcm2, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| expected | rank sum | obs | grupo |
|------------|------------|----------|------------------|
| 825<br>660 | 858<br>627 | 30<br>24 | MEP <br>CONTROL |
| 1485 | 1485 | <br>54 | combined |

unadjusted variance 3300.00 adjustment for ties -4.91 ------ adjusted variance 3295.09

Ho: updpos $\sim$ 2(grupo==MEP) = updpos $\sim$ 2(grupo==CONTROL) z = 0.575

Prob > |z| = 0.5654

. ranksum upd2kgcm2, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| grupo | obs | rank sum | expected |
|------------------|----------|------------|------------|
| MEP <br>CONTROL | 30<br>24 | 937<br>548 | 825<br>660 |
| combined | <br>54 | 1485 | 1485 |

unadjusted variance 3300.00

adjustment for ties -6.42

-----

adjusted variance 3293.58

Ho: upd2kg~2(grupo==MEP) = upd2kg~2(grupo==CONTROL)

z = 1.952

Prob > |z| = 0.0510

. ranksum updda3kgcm2, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| expected | rank sum | obs | grupo |
|------------|------------|----------|------------------|
| 825<br>660 | 927<br>558 | 30<br>24 | MEP <br>CONTROL |
| 1485 | 1485 | <br>54 | |

unadjusted variance 3300.00

adjustment for ties -6.92

adjusted variance 3293.08

Ho: updda3~2(grupo==MEP) = updda3~2(grupo==CONTROL)

z = 1.777

Prob > |z| = 0.0755

. ranksum DELTAUPDPREPOST, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| expected | rank sum | obs | grupo |
|------------|------------|----------|------------------|
| 825<br>660 | 847<br>638 | 30<br>24 | MEP <br>CONTROL |
| 1485 | 1485 | 54 | combined |

unadjusted variance 3300.00

adjustment for ties -1.76

adjusted variance 3298.24

Ho: DELTAU~T(grupo==MEP) = DELTAU~T(grupo==CONTROL) 
$$z = 0.383$$
 
$$Prob > |z| = 0.7017$$

#### . ranksum DELTAUPDDOSPRE, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| grupo | obs | rank sum | expected |
|----------------|-----|------------|------------|
| MEP<br>CONTROL | | 897<br>588 | 825<br>660 |
| combined | 54 | <br>1485 | 1485 |

unadjusted variance 3300.00 adjustment for ties -2.64 -------- adjusted variance 3297.36

Ho: DELTAU..(grupo==MEP) = DELTAU..(grupo==CONTROL) 
$$z = 1.254$$
 
$$Prob > |z| = 0.2099$$

#### . ranksum DELTAUPDTRESPRE, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| expected | rank sum | obs | grupo |
|------------|------------|----------|------------------|
| 825<br>660 | 859<br>626 | 30<br>24 | MEP <br>CONTROL |
| 1485 | 1485 | +54 | combined |

unadjusted variance 3300.00 adjustment for ties -0.63 ------ adjusted variance 3299.37

Ho: DELTAU..(grupo==MEP) = DELTAU..(grupo==CONTROL)  

$$z = 0.592$$

Prob > |z| = 0.5539

. bysort grupo:swilk idprelevamm idpostlevamm id2evamm idda3evamm DELTAIDPOSTPRE DELTAIDDOSPRE DELTAIDTRESPRE

-----

-----

-> grupo = MEP

Shapiro-Wilk W test for normal data

| Variable | Obs | W | V | Z | Prob>z |
|--------------|-----|---------|-------|-------|---------|
| idpre1evamm | 30 | 0.95125 | 1.550 | 0.906 | 0.18256 |
| idpost1evamm | 30 | 0.94528 | 1.739 | 1.144 | 0.12625 |
| id2evamm | 30 | 0.96659 | 1.062 | 0.125 | 0.45045 |
| idda3evamm | 30 | 0.94067 | 1.886 | 1.312 | 0.09480 |
| DELTAIDPOS~E | 30 | 0.96762 | 1.029 | 0.059 | 0.47640 |
| DELTAIDDOS~E | 30 | 0.90787 | 2.928 | 2.222 | 0.01315 |
| DELTAIDTRE~E | 30 | 0.96509 | 1.110 | 0.215 | 0.41481 |

\_\_\_\_\_\_

-----

Shapiro-Wilk W test for normal data

| Variable | Obs | W | V | Z | Prob>z |
|--------------|-----|---------|-------|--------|---------|
| | + | | | | |
| idpre1evamm | 24 | 0.97700 | 0.620 | -0.974 | 0.83489 |
| idpost1evamm | 24 | 0.96140 | 1.041 | 0.082 | 0.46713 |
| id2evamm | 24 | 0.96554 | 0.929 | -0.149 | 0.55932 |
| idda3evamm | 24 | 0.90705 | 2.507 | 1.874 | 0.03045 |
| DELTAIDPOS~E | 24 | 0.97590 | 0.650 | -0.878 | 0.81008 |
| DELTAIDDOS~E | 24 | 0.81556 | 4.975 | 3.271 | 0.00054 |
| DELTAIDTRE~E | 24 | 0.92705 | 1.968 | 1.380 | 0.08376 |

. bysort grupo:sum idprelevamm idpostlevamm id2evamm idda3evamm DELTAIDPOSTPRE DELTAIDDOSPRE DELTAIDTRESPRE, detail

\_\_\_\_\_

-----

<sup>-&</sup>gt; grupo = CONTROL

<sup>-&</sup>gt; grupo = MEP

ID PRE 1 (EVA. mm)

| | | · | | |
|-----|-------------|-----------------|-------------|----------|
| | Percentiles | Smallest | | |
| 1% | 12 | 12 | | |
| 5% | 12 | 12 | | |
| 10% | 15 | 15 | Obs | 30 |
| 25% | 21 | 15 | Sum of Wgt. | 30 |
| 50% | 32 | | Mean | 33.6 |
| | | Largest | Std. Dev. | 13.79555 |
| 75% | 47 | 49 | | |
| 90% | 50 | 51 | Variance | 190.3172 |
| 95% | 51 | 51 | Skewness | 0221884 |
| 99% | 60 | 60 | Kurtosis | 1.854865 |
| | | ID POST 1 (EVA. | mm) | |
| | Percentiles | Smallest | | |
| 1% | 7 | 7 | | |
| 5% | 7 | 7 | | |
| 10% | 9.5 | 8 | 0bs | 30 |
| 25% | 15 | 11 | Sum of Wgt. | 30 |
| 50% | 23.5 | | Mean | 25.03333 |
| | | Largest | Std. Dev. | 12.20086 |
| 75% | 38 | 40 | | |
| 90% | 40.5 | 41 | Variance | 148.8609 |
| 95% | 43 | 43 | Skewness | .1581778 |
| 99% | 48 | 48 | Kurtosis | 1.760058 |
| | | ID 2 (EVA. mm | ) | |
| | Percentiles | Smallest | | |
| 1% | 7 | 7 | | |
| 5% | 8 | 8 | | |
| 10% | 9 | 8 | 0bs | 30 |
| 25% | 14 | 10 | Sum of Wgt. | 30 |
| | | | - | |
| 50% | 21 | | Mean | 22.73333 |
| | | Largest | Std. Dev. | 10.88793 |
| 75% | 30 | 36 | | |
| 90% | 38 | 40 | Variance | 118.5471 |

| 95%<br>99% | 45<br>45 | 45<br>45 | Skewness<br>Kurtosis | .4615728<br>2.28832 |
|---|---|---|---|---|
| | | ID día 3 (EVA. | . mm) | |
| | Percentiles | <br>Smallest | | |
| 1% | 5 | 5 | | |
| 5% | 5 | 5 | | |
| 10% | 6.5 | 5 | Obs | 30 |
| 25% | 10 | 8 | Sum of Wgt. | 30 |
| 50% | 19.5 | | Mean | 18.96667 |
| | | Largest | Std. Dev. | 9.96713 |
| 75% | 28 | 30 | | 2.00. |
| 90% | 30 | 30 | Variance | 99.34368 |
| 95% | 35 | 35 | Skewness | .20909 |
| 99% | 40 | 40 | Kurtosis | 1.904974 |
| | | DELTAIDPOST | PRE | |
| | Percentiles | Smallest | | |
| 1% | -23 | -23 | | |
| 5% | -22 | -22 | | |
| 10% | -17.5 | -18 | Obs | 30 |
| 25% | -14 | -17 | Sum of Wgt. | 30 |
| 50% | -9 | | Mean | -8.566667 |
| | | Largest | Std. Dev. | 8.173478 |
| 75% | -5 | -1 | | |
| 90% | .5 | 2 | Variance | 66.80575 |
| 95% | 10 | 10 | Skewness | .6031255 |
| 99% | 12 | 12 | Kurtosis | 3.372561 |
| | | DELTAIDDOSF | PRE | |
| | Percentiles | Smallest | | |
| 1% | -30 | -30 | | |
| 5% | -26 | -26 | | |
| 10% | -22 | -22 | Obs | 30 |
| 25% | -18 | -22 | Sum of Wgt. | 30 |
| 50% | -14 | | Mean | -10.86667 |
| | | Largest | Std. Dev. | 11.49433 |

| 75% | -5 | 2 | | |
|-----|----|----|----------|----------|
| 90% | 3 | 4 | Variance | 132.1195 |
| 95% | 10 | 10 | Skewness | 1.35135 |
| 99% | 28 | 28 | Kurtosis | 5.713002 |

#### DELTAIDTRESPRE

| | Percentiles | Smallest | | |
|-----|-------------|----------|-------------|-----------|
| 1% | -33 | -33 | | |
| 5% | -31 | -31 | | |
| 10% | -30.5 | -31 | Obs | 30 |
| 25% | -24 | -30 | Sum of Wgt. | 30 |
| 50% | -15 | | Mean | -14.63333 |
| | | Largest | Std. Dev. | 11.7927 |
| 75% | -9 | 1 | | |
| 90% | 1.5 | 2 | Variance | 139.0678 |
| 95% | 5 | 5 | Skewness | .5150803 |
| 99% | 17 | 17 | Kurtosis | 3.165103 |

\_\_\_\_\_

-----

## ID PRE 1 (EVA. mm)

| | Percentiles | Smallest | | |
|-----|-------------|----------------|-------------|----------|
| 1% | 6 | 6 | | |
| 5% | 7 | 7 | | |
| 10% | 10 | 10 | Obs | 24 |
| 25% | 20.5 | 13 | Sum of Wgt. | 24 |
| 50% | 29.5 | | Mean | 31.41667 |
| | | Largest | Std. Dev. | 15.10519 |
| 75% | 40 | 48 | | |
| 90% | 49 | 49 | Variance | 228.1667 |
| 95% | 59 | 59 | Skewness | .1359331 |
| 99% | 61 | 61 | Kurtosis | 2.376209 |
| | | TD BOST 1 (EVA | mm) | |

#### ID POST 1 (EVA. mm)

-----

Percentiles Smallest 1% 2 2

<sup>-&</sup>gt; grupo = CONTROL

| 5% | 3 | 3 | | |
|-----|-------------|------------------|-------------|-----------|
| 10% | 9 | 9 | Obs | 24 |
| 25% | 13.5 | 10 | Sum of Wgt. | 24 |
| | | | - | |
| 50% | 23 | | Mean | 24.83333 |
| | | Largest | Std. Dev. | 15.11598 |
| 75% | 33.5 | 42 | | |
| 90% | 48 | 48 | Variance | 228.4928 |
| 95% | 52 | 52 | Skewness | . 5737374 |
| 99% | 59 | 59 | Kurtosis | 2.644348 |
| | | ID 2 (EVA. mm) | ) | |
| | Percentiles | Smallest | | |
| 1% | 3 | 3 | | |
| 5% | 3 | 3 | | |
| 10% | 6 | 6 | Obs | 24 |
| 25% | 12 | 8 | Sum of Wgt. | 24 |
| 50% | 24 | | Mean | 23.83333 |
| | | Largest | Std. Dev. | 14.01138 |
| 75% | 32.5 | 35 | | |
| 90% | 40 | 40 | Variance | 196.3188 |
| 95% | 45 | 45 | Skewness | .5143827 |
| 99% | 60 | 60 | Kurtosis | 3.103797 |
| | | ID día 3 (EVA. r | nm) | |
| | Percentiles | Smallest | | |
| 1% | | 3 | | |
| 5% | 3 | 3 | | |
| 10% | 4 | 4 | Obs | 24 |
| 25% | 10.5 | 6 | Sum of Wgt. | 24 |
| 50% | 18.5 | | Mean | 19.95833 |
| | | Largest | Std. Dev. | 13.22869 |
| 75% | 25.5 | 34 | | |
| 90% | 34 | 34 | Variance | 174.9982 |
| 95% | 41 | 41 | Skewness | 1.162349 |
| 99% | 60 | 60 | Kurtosis | 4.691994 |
| | | DELTAIDPOSTPRE | Ē | |

| | Percentiles | Smallest | | |
|---|---|---|---|---|
| 1% | -29 | -29 | | |
| 5% | -16 | -16 | | |
| 10% | -15 | -15 | Obs | 24 |
| 25% | -11.5 | -15 | Sum of Wgt. | 24 |
| F.00/ | 7 | | Mass | C |
| 50% | -7 | Lamasat | Mean | -6.583333 |
| 7.50/ | F | Largest | Std. Dev. | 8.632178 |
| 75% | 5 | 2 | Vaniana | 74 51440 |
| 90% | 3<br>7 | 3 | Variance | 74.51449 |
| 95%<br>99% | ,<br>11 | 7<br>11 | Skewness<br>Kurtosis | 260452<br>3.466838 |
| 99/0 | 11 | 11 | Kui tos is | 3.400030 |
| | | DELTAIDDOSF | PRE | |
| | Percentiles | Smallest | | |
| 1% | -21 | -21 | | |
| 5% | -19 | -19 | | |
| 10% | -18 | -18 | Obs | 24 |
| 25% | -15 | -18 | Sum of Wgt. | 24 |
| 50% | -10.5 | | Mean | -7.583333 |
| | | Largest | Std. Dev. | 12.1115 |
| 75% | -4.5 | 2 | | |
| 90% | 7 | 7 | Variance | 146.6884 |
| 95% | 13 | 13 | Skewness | 1.905437 |
| 99% | 34 | 34 | Kurtosis | 6.987127 |
| | | DELTAIDTRES | PRE | |
| | Percentiles | Smallest | | |
| 1% | -28 | -28 | | |
| 5% | -27 | -27 | | |
| 10% | -26 | -26 | Obs | 24 |
| 25% | -21.5 | -26 | Sum of Wgt. | 24 |
| | | | J | |
| 50% | -14 | | Mean | -11.45833 |
| | | Largest | Std. Dev. | 13.11812 |
| 75% | -3 | -1 | | |
| 90% | 9 | 9 | Variance | 172.0851 |
| 95% | 15 | 15 | Skewness | .8250901 |
| 99% | 20 | 20 | Kurtosis | 2.989924 |

```
. bysort grupo:tabstat idprelevamm, s(med iqr)
-> grupo = MEP
 variable | p50 iqr
-----
         32
idpre1evamm |
_____
______
-> grupo = CONTROL
 variable | p50 iqr
-----
idprelevamm | 29.5
. bysort grupo:tabstat idprelevamm, s(med p25 p75)
-> grupo = MEP
 variable | p50 p25
 -----
idprelevamm | 32 21
                    47
 -----
-> grupo = CONTROL
  variable | p50 p25 p75
 -----
idprelevamm | 29.5 20.5
```

. ranksum idprelevamm, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| grupo | obs | rank sum | expected |
|------------------|----------|------------|------------|
| MEP <br>CONTROL | 30<br>24 | 865<br>620 | 825<br>660 |
| combined | 54 | 1485 | 1485 |

unadjusted variance 3300.00
adjustment for ties -5.41
----adjusted variance 3294.59

Ho: idpre1~m(grupo==MEP) = idpre1~m(grupo==CONTROL) z = 0.697 Prob > |z| = 0.4859

. ranksum idpost1evamm, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| expected | rank sum | l obs | grupo |
|------------|------------|-----------|----------------|
| 825<br>660 | 837<br>648 | • | MEP<br>CONTROL |
| 1485 | 1485 | +<br> 54 | combined |

unadjusted variance 3300.00
adjustment for ties -7.04
----adjusted variance 3292.96

Ho: idpost~m(grupo==MEP) = idpost~m(grupo==CONTROL) z = 0.209 Prob > |z| = 0.8344

. ranksum id2evamm, by(grupo)

Two-sample wilcoxon rank-sum (Mann-whitney) test

grupo | obs rank sum expected

| | -+ | | |
|----------|-----------|------|------|
| MEP | 30 | 814 | 825 |
| CONTROL | 24 | 671 | 660 |
| combined | +<br> 54 | 1485 | 1485 |

unadjusted variance
adjustment for ties
-6.79
----adjusted variance
3300.00
----3293.21

Ho: id2evamm(grupo==MEP) = id2evamm(grupo==CONTROL) z = -0.192Prob > |z| = 0.8480

. ranksum idda3evamm, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| expected | rank sum | obs | grupo |
|------------|------------|-----------|----------------|
| 825<br>660 | 832<br>653 | | MEP<br>CONTROL |
| 1485 | 1485 | +<br> 54 | combined |

unadjusted variance 3300.00 adjustment for ties -7.17 ------ adjusted variance 3292.83

Ho: idda3e~m(grupo==MEP) = idda3e~m(grupo==CONTROL) z = 0.122 Prob > |z| = 0.9029

. ranksum DELTAIDPOSTPRE, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| grupo | obs | rank sum | expected |
|---------|-----|----------|----------|
| MEP | 30 | 759.5 | 825 |
| CONTROL | 24 | 725.5 | 660 |

unadjusted variance 3300.00 adjustment for ties -10.69

-----

adjusted variance 3289.31

Ho: DEL~TPRE(grupo==MEP) = DEL~TPRE(grupo==CONTROL)

z = -1.142

Prob > |z| = 0.2534

. ranksum DELTAIDDOSPRE, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| rank sum expected | obs | grupo |
|----------------------|----------|------------------|
| 759.5 82<br>725.5 66 | 30<br>24 | MEP <br>CONTROL |
| 723.3 00<br>1485 148 | <br>54 | complined |

unadjusted variance 3300.00 adjustment for ties -10.57

adjusted variance 3289.43

Ho: DELTAI..(grupo==MEP) = DELTAI..(grupo==CONTROL)

z = -1.142

Prob > |z| = 0.2534

. ranksum DELTAIDTRESPRE, by(grupo)

Two-sample Wilcoxon rank-sum (Mann-Whitney) test

| grupo | l obs | rank sum | expected |
|----------|-------|----------|----------|
| | + | | |
| MEP | 30 | 786 | 825 |
| CONTROL | 24 | 699 | 660 |
| | + | | |
| combined | 54 | 1485 | 1485 |

```
unadjusted variance 3300.00 adjustment for ties -6.29 ------adjusted variance 3293.71
```

Ho: DELTAI..(grupo==MEP) = DELTAI..(grupo==CONTROL) z = -0.680 Prob > |z| = 0.4968

- . h constant comparative
- . gen UPD11MEP=.
  (54 missing values generated)
- . replace UPD11MEP= DELTAUPDPREPOST if grupo==1
  (30 real changes made)
- . drop UPD11MEP
- . gen UPDPREMEP=.
  (54 missing values generated)
- . gen UPDPREMEP= updpre1kgcm2 if grupo==1
  UPDPREMEP already defined
  r(110);
- . replace UPDPREMEP= updpre1kgcm2 if grupo==1
  (30 real changes made)
- . gen UPDPOSTMEP= updpost1kgcm2 if grupo==1
  (24 missing values generated)
- . gen UPD2MEP= upd2kgcm2 if grupo==1
  (24 missing values generated)
- . gen UPD3MEP = updda3kgcm2 if grupo==1
  (24 missing values generated)
- . by(grupo):signrank DELTAUPDPREPOST
  invalid syntax
  r(198);
- . h signrank

#### . signrank updpre1kgcm2= updpost1kgcm2

### Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 7 | 131.5 | 741 |
| negative | 45 | 1350.5 | 741 |
| zero | 2 | 3 | 3 |
| + | | | |
| all | 54 | 1485 | 1485 |

unadjusted variance 13488.75
adjustment for ties -2.00
adjustment for zeros -1.25
----adjusted variance 13485.50

Ho: updpre1kgcm2 = updpost1kgcm2

z = -5.249Prob > |z| = 0.0000

. signrank UPDPREMEP= UPDPOSTMEP

#### Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|--------|-----------|----------|
| positive | 5 | 54 | 232.5 |
| negative | 25 | 411 | 232.5 |
| zero | 0 | 0 | 0 |
| all | <br>30 | 465 | 465 |

unadjusted variance 2363.75
adjustment for ties -0.25
adjustment for zeros 0.00
-----adjusted variance 2363.50

Ho: UPDPREMEP = UPDPOSTMEP z = -3.672

Prob > |z| = 0.0002

. bysort grupo:signrank updpre1kgcm2= updpost1kgcm2

-----

-----

-> grupo = MEP

Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 5 | 54 | 232.5 |
| negative | 25 | 411 | 232.5 |
| zero | 0 | 0 | 0 |
| all | 30 | 465 | 465 |

unadjusted variance 2363.75
adjustment for ties -0.25
adjustment for zeros 0.00
----adjusted variance 2363.50

Ho: updpre1kgcm2 = updpost1kgcm2

z = -3.672

Prob > |z| = 0.0002

-----

-----

-> grupo = CONTROL

Wilcoxon signed-rank test

| sum ranks | obs | sign |
|-----------|-----------|-----------------------|
| 15 | 2 | positive |
| 282 | 20 | negative |
| 3 | 2 | zero |
| 300 | 24 | all |
| | 15<br>282 | 2 15<br>20 282<br>2 3 |

unadjusted variance 1225.00

adjustment for ties -0.12 adjustment for zeros -1.25 adjusted variance 1223.62 Ho: updpre1kgcm2 = updpost1kgcm2 z = -3.816Prob > |z| = 0.0001. bysort grupo:tabstat DELTAUPDPREPOST, s(med p25 p75) \_\_\_\_\_ -> grupo = MEP variable | p50 p25 p75 -----DELTAUPDPR~T | .17 .0500001 \_\_\_\_\_ -> grupo = CONTROL variable | p50 p25 p75 -----DELTAUPDPR~T | .135 .045 .265 . bysort grupo:signrank updpre1kgcm2= upd2kgcm2 -> grupo = MEP Wilcovon signed-rank tost

| WΙ | rcoxon | Signed-rank | test |
|----|--------|-------------|------|

| sign | l obs | sum ranks | expected |
|----------|-------|-----------|----------|
| positive | -+4 | 13 | 232.5 |
| negative | 26 | 452 | 232.5 |
| zero | 0 | 0 | 0 |
| | -+ | | |

all | 30 465 465

unadjusted variance 2363.75
adjustment for ties -0.38
adjustment for zeros 0.00

adjusted variance 2363.38

Ho: updpre1kgcm2 = upd2kgcm2

z = -4.515

Prob > |z| = 0.0000

-----

-----

-> grupo = CONTROL

Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 2 | 16 | 150 |
| negative | 22 | 284 | 150 |
| zero | 0 | 0 | 0 |
| +- | | | |
| all | 24 | 300 | 300 |

unadjusted variance 1225.00 adjustment for ties -0.25 adjustment for zeros 0.00

adjusted variance 1224.75

Ho: updpre1kgcm2 = upd2kgcm2

z = -3.829

Prob > |z| = 0.0001

. bysort grupo:tabstat DELTAUPDDOSPRE, s(med p25 p75)

-----

-----

-> grupo = MEP

variable | p50 p25 p75

DELTAUPDDO~E | .3 .1 .4899999

-> grupo = CONTROL

| variable | p25 | p75 |
|--------------|------|-----|
| DELTAUPDDO~E | .105 | .29 |

. bysort grupo:signrank updpre1kgcm2=updda3kgcm2

\_\_\_\_\_

-----

-> grupo = MEP

Wilcoxon signed-rank test

| expected | sum ranks | obs | sign |
|----------|-----------|-----|----------|
| 232.5 | 0 | 0 | positive |
| 232.5 | 465 | 30 | negative |
| 0 | 0 | 0 | zero |
| | | + | |
| 465 | 465 | 30 | all |

unadjusted variance 2363.75
adjustment for ties -0.25
adjustment for zeros 0.00
-----adjusted variance 2363.50

Ho: updpre1kgcm2 = updda3kgcm2

z = -4.782

Prob > |z| = 0.0000

-----

-----

-> grupo = CONTROL

37

#### Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 3 | 14 | 149.5 |
| negative | 20 | 285 | 149.5 |
| zero | 1 | 1 | 1 |
| all | 24 | 300 | 300 |

unadjusted variance 1225.00 adjustment for ties -0.12 adjustment for zeros -0.25 ------- adjusted variance 1224.62

Ho: updpre1kgcm2 = updda3kgcm2 z = -3.872Prob > |z| = 0.0001

. bysort grupo:tabstat DELTAUPDTRESPRE, s(med p25 p75)

-----

-> grupo = MEP

| variable | p50 | p25 | p75 |
|--------------|------|-----|-----|
| DELTAUPDTR~E | .335 | .13 | .52 |

\_\_\_\_\_

\_\_\_\_\_

-----

-> grupo = CONTROL

| variable | • | p25 | p75 |
|--------------|---|------|-----|
| DELTAUPDTR~E | | .145 | .43 |

. by sort grupo:signrank idprelevamm= idpostlevamm -----

\_\_\_\_\_

-> grupo = MEP

Wilcoxon signed-rank test

| sign | | obs | sum ranks | expected |
|----------|---|-----|-----------|----------|
| positive | | 27 | 426 | 232.5 |
| negative | | 3 | 39 | 232.5 |
| zero | | 0 | 0 | 0 |
| | + | | | |
| all | 1 | 30 | 465 | 465 |

unadjusted variance 2363.75
adjustment for ties -2.62
adjustment for zeros 0.00
-----adjusted variance 2361.12

Ho: idpre1evamm = idpost1evamm

z = 3.982

Prob > |z| = 0.0001

-----

-----

-> grupo = CONTROL

Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 18 | 258 | 148.5 |
| negative | 4 | 39 | 148.5 |
| zero | 2 | 3 | 3 |
| + | | | |
| all | 24 | 300 | 300 |

unadjusted variance 1225.00 adjustment for ties -1.25 adjustment for zeros -1.25 ------adjusted variance 1222.50

```
Ho: idpre1evamm = idpost1evamm
       z = 3.132
  Prob > |z| = 0.0017
. bysort grupo:tabstat DELTAIDPOSTPRE, s(med p25 p75)
-> grupo = MEP
  variable | p50 p25 p75
-----
DELTAIDPOS~E |
           -9
                 -14
-> grupo = CONTROL
  variable | p50 p25 p75
-----
DELTAIDPOS~E |
           -7 -11.5 -.5
. bysort grupo:tabstat DELTAIDDOSPRE, s(med p25 p75)
-> grupo = MEP
  variable | p50 p25 p75
-----
            -14
                  -18
DELTAIDDOS~E |
_____
-----
-> grupo = CONTROL
  variable | p50 p25 p75
```

-4.5

-15

DELTAIDDOS~E | -10.5

. bysort grupo:tabstat DELTAIDTRESPRE, s(med p25 p75)

\_\_\_\_\_

-----

-> grupo = MEP

| variable | • | p25 | p75 |
|--------------|---|-----|-----|
| DELTAIDTRE~E | | -24 | -9 |

-----

-----

-> grupo = CONTROL

| variable | p50 | p25 | p75 |
|--------------|-----|-------|-----|
| DELTAIDTRE~E | | -21.5 | -3 |

. bysort grupo:signrank idprelevamm= id2evamm

\_\_\_\_\_

-----

-> grupo = MEP

Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 26 | 421 | 232.5 |
| negative | 4 | 44 | 232.5 |
| zero | 0 | 0 | 0 |
| | -+ | | |
| all | 30 | 465 | 465 |

unadjusted variance 2363.75
adjustment for ties -2.62
adjustment for zeros 0.00
-----adjusted variance 2361.12

Ho: idpre1evamm = id2evamm  

$$z = 3.879$$
  
Prob >  $|z| = 0.0001$ 

-----

\_\_\_\_\_

-> grupo = CONTROL

Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 20 | 255 | 150 |
| negative | 4 | 45 | 150 |
| zero | 0 | 0 | 0 |
| + | | | |
| all | 24 | 300 | 300 |

unadjusted variance 1225.00 adjustment for ties -2.12 adjustment for zeros 0.00 ------adjusted variance 1222.88

Ho: idprelevamm = id2evamm z = 3.003

Prob > |z| = 0.0027

. bysort grupo:signrank idprelevamm= idda3evamm

-----

-----

-> grupo = MEP

Wilcoxon signed-rank test

| sign | | obs | sum ranks | expected |
|----------|------|-----|-----------|----------|
| positive | • | 26 | 440.5 | 232.5 |
| negative | | 4 | 24.5 | 232.5 |
| zero | <br> | 0 | 0 | 0 |

| all | 30 | 465 | 465 |
|-----|----|-----|-----|
| α | 30 | 103 | 103 |

unadjusted variance 2363.75
adjustment for ties -1.25
adjustment for zeros 0.00
-----adjusted variance 2362.50

Ho: idprelevamm = idda3evamm

z = 4.279

Prob > |z| = 0.0000

-----

-----

-> grupo = CONTROL

Wilcoxon signed-rank test

| sign | obs | sum ranks | expected |
|----------|-----|-----------|----------|
| positive | 21 | 264.5 | 150 |
| negative | 3 | 35.5 | 150 |
| zero | 0 | 0 | 0 |
| all | 24 | 300 | 300 |

unadjusted variance 1225.00 adjustment for ties -1.12 adjustment for zeros 0.00 -------adjusted variance 1223.88

Ho: idpre1evamm = idda3evamm

z = 3.273

Prob > |z| = 0.0011

- . graph box DELTAUPDPREPOST DELTAUPDDOSPRE DELTAUPDTRESPRE, over(grupo)
- . bysort grupo:swilk distanciapec7cruzcm

-----

-----

-> grupo = MEP

# Shapiro-Wilk W test for normal data

| Variable <br> | | | | z | Prob>z |
|---|---|---|---|---|---|
| distanciap~m | | | | 3.651 | 0.00013 |
| -> grupo = CONTROL | | | | | |
| Shapiro-Wilk W test for normal data | | | | | |
| Variable | | | | | |
| distanciap~m | | | | | |
| . bysort grupo:tabstat distanciapec7cruzcm, s(med p25 p75) | | | | | |
| -> grupo = MEP | | | _ | | |
| variable <br>+ | | | | | |
| distanciap~m | 8.6 | | 9.5 | | |
| | | | - | | |
| -> grupo = CONTRO | | 25 | <b>7</b> 5 | | |
| variable <br>+ | | | | | |
| distanciap~m | | | | | |
| . ranksum distanciapec7cruzcm, by( grupo) | | | | | |
| Two-sample Wilcoxon rank-sum (Mann-Whitney) test | | | | | |
| grupo obs rank sum expected | | | | | |

| MEP | 30 | 856 | 825 |
|----------|----|------|------|
| CONTROL | 24 | 629 | 660 |
| + | | | |
| combined | 54 | 1485 | 1485 |

unadjusted variance
adjustment for ties
-12.20
----adjusted variance
3300.00
-12.20
----3287.80

Ho: distan~m(grupo==MEP) = distan~m(grupo==CONTROL) z = 0.541

Prob > |z| = 0.5888

.